CLINICAL TRIAL: NCT05723679
Title: Targeting Breathing Limitations to Improve Functional Outcomes in Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Targeting Breathing Limitations to Improve Functional Outcomes in HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Bryce Balmain, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STU-2022-1174
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Obesity
Keywords: exertional dyspnea; exercise intolerance; HFpEF; breathing limitations; cardiopulmonary physiology
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Mechanistic Clinical Trial
Who Masked: Participant
Masking Description: The order of the room air and HeO2 tests will be randomized and the subjects will not be told what gas mixture they will be breathing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeO2 gas mixture, then Room air gas mixture (Experimental): Participant will be randomized to each intervention on separate days (Study visit 3 and 4) in this cross-over trial. Participants that receive HeO2 first will then receive the room air gas mixture. At least 24 hours will separate each visit.
  Interventions: Other: HeO2 gas mixture; Other: Room air gas mixture
- Room air gas mixture, then HeO2 gas mixture (Experimental): Participant will be randomized to each intervention on separate days (Study visit 3 and 4) in this cross-over trial. Participants that receive Room air first will then receive the HeO2 mixture. At least 24 hours will separate each visit.
  Interventions: Other: HeO2 gas mixture; Other: Room air gas mixture

INTERVENTIONS:
Other: HeO2 gas mixture — Low-density helium-oxygen gas mixture (HeO2: 21% O2 and 79% He). Participant will be breathing this gas mixture.
Other: Room air gas mixture — Normal room air

SUMMARY:
The overall purpose of this study is to investigate whether pulmonary limitations that increase the oxygen (O2) cost of breathing impact dyspnea on exertion (DOE) and peak exercise capacity in patients with HFpEF and obesity. As per investigator's hypothesis, obesity is likely a significant contributor to DOE and exercise intolerance in patients with HFpEF.

DETAILED DESCRIPTION:
Clinical screening tests including cardiopulmonary exercise testing (CPET), pulmonary function testing, and dual-energy x-ray absorptiometry (DEXA) scans will be performed on all subjects. Investigator's approach will be to undertake the following objectives:

Objective 1: (Observational) is a cross-sectional study designed to test the interaction of HFpEF (underlying changes in pulmonary function) and obesity (obesity-related changes in pulmonary function) on the O2 cost of breathing, and its association with DOE and peak exercise capacity. The specific hypotheses proposed to test as part of this objective are:

Hypothesis 1.1: Due to the presence of obesity-related mechanical ventilatory constraints, the O2 cost of breathing will be greater in obese HFpEF patients and obese controls vs. nonobese HFpEF patients and nonobese controls, but will be similar between obese HFpEF patients vs. obese controls.

Hypothesis 1.2: The association between the O2 cost of breathing and DOE and the association between the O2 cost of breathing and peak exercise capacity will be stronger in obese HFpEF patients and obese controls vs. nonobese HFpEF patients and nonobese controls, but will be similar between obese HFpEF patients vs. obese controls.

Objective 2: (Interventional) is a single-blind, randomized, placebo-controlled, cross-over trial designed to investigate the effects of reducing obesity-related mechanical ventilatory constraints by breathing a HeO2 gas mixture (HeO2: 21% O2 and 79% He) on DOE and peak exercise capacity. The specific hypotheses proposed to test as part of this objective are:

Hypothesis 2.1: HeO2 will decrease DOE in obese HFpEF patients and obese controls, but not in nonobese HFpEF patients or nonobese controls, as HFpEF- or cardiovascular-related limitations will not be affected by HeO2.

Hypothesis 2.2: HeO2 will increase peak exercise capacity in obese HFpEF patients and obese controls, but not in nonobese HFpEF patients or nonobese controls as HFpEF- or cardiovascular-related limitations will not be affected by HeO2.

Study Day 1:

This visit consists of a consenting process (including medical Hx , DEXA scan, and pulmonary function testing. Goals of this day are to determine fat and lean mass and to quantify pulmonary function. This visit will usually last between 3 - 3.5 hours. Any subjects who demonstrate severe pulmonary disease at this point will be excluded.

Study Day 2:

This visit will consist of O2 cost of breathing tests, as well as submaximal and maximal CPET tests. This visit is designed to test Hypotheses 1.1 and 1.2. and will usually last between 3 - 3.5 hours.

Study Day 3 and 4:

These visits consist of submaximal and maximal CPET tests with either breathing room air or HeO2 gas mixtures on separate days. These visits are designed to test Hypotheses 2.1 and 2.2. and will usually last between 2 - 2.5 hours.

The Diagnostic test including : 1) Submaximal and maximal cardiopulmonary exercise test 2) pulmonary function testing 3) Eucapnic Voluntary Hyperventilation 3) Dual-Energy X-Ray absorptiometry (DEXA), are the procedures that will be performed by the participants for investigator to gather data (observational) and assess DOE, peak exercise capacity, pulmonary function, body composition, and O2 cost of breathing between study groups.

ELIGIBILITY:
Inclusion Criteria:

* signs and symptoms of heart failure
* an ejection fraction > 0.50;
* objective evidence of diastolic dysfunction. elevated biomarkers (NT-proBNP >300 ng/dl) or HF hospitalization
* healthy volunteers

Exclusion Criteria:

* age < 55 years
* BMI > 50 kg/m2
* Atrial fibrillation with poorly controlled heart rate
* phosphodiesterase type 5 (PDE5) inhibitor use
* severe valvular disease
* severe Chronic obstructive pulmonary disease (COPD)
* Chronic kidney disease (CKD) 4 or higher
* any restriction of ambulation and mobility.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
O2 cost of breathing (Objective 1) | Day 2
  O2 cost of breathing measured during eucapnic voluntary hyperventilation, and calculated using oxygen uptake and ventilation variables.
Change in DOE during HeO2 breathing (Objective 2) | Day 3 or 4
  Dyspnea on Exertion (DOE) will be assessed via ratings of perceived breathlessness (RPB) using a 0-10 Borg Scale, and will be compared with that measured during room air breathing.
Change in peak exercise capacity during HeO2 breathing (Objective 2) | Day 3 or 4
  Peak exercise capacity will be assessed by measuring peak oxygen uptake (in L/min, measured via a breath-by-breath metabolic measurement system), peak power output recorded from a cycle ergometer (Watts), and/or total exercise duration (minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Tony G Babb, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center; Bryce N Balmain, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No